CLINICAL TRIAL: NCT06779903
Title: Effect Of Psychoeducatıon Interventıon For Postpartum Care On Postpartum Depressıon And Breastfeedıng
Brief Title: Psychoeducatıon Interventıon Postpartum Depressıon Breastfeedıng
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Yasemin Ozhuner, Principal Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSYCHOEDUCATION DEPRESSION
Record Dates: First submitted 2024-12-11; First posted 2025-01-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Depression; Psychoeducation; Breastfeeding; Postpartum Care
Keywords: Postpartum depression; Watson model; psychoeducation; breastfeeding
MeSH Terms: conditions — Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Intervention Model Description: The pregnant women included in the sample were informed about the study and their written informed consent was obtained. Six interviews were conducted with the pregnant women, four at one-week intervals before birth, and one on the tenth day and sixth week after birth. These interviews were conducted with the women one-on-one and face-to-face.Women in the control group were not given any treatment other than routine care at family health centers. The psychoeducation program was applied to the women in the intervention group in six interviews.
Who Masked: Participant
Masking Description: control group (55) intervention group (55)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The pregnant women included in the sample were informed about the study and their written informed consent was obtained. Six interviews were conducted with the pregnant women, four at one-week intervals before birth, and one on the tenth day and sixth week after birth. These interviews were conducted with the women one-on-one and face-to-face. psychoeducation program was applied to the women in the intervention group in six interviews.In the first interview, the psychoeducation intervention program booklet based on the Watson Model for postpartum care was given to the women and the interview was conducted within the scope of the program. The psychoeducation intervention program sessions based on the Watson Model for postpartum care in the study were conducted according to the WİBM improvement processes and psychoeducation techniques. The interviews lasted between 90 and 120 minutes on average.
  Interventions: Other: the psychoeducation intervention program booklet
- control group (Placebo Comparator): The pregnant women included in the sample were informed about the study and their written informed consent was obtained. Six interviews were conducted with the pregnant women, four at one-week intervals before birth, and one on the tenth day and sixth week after birth. These interviews were conducted with the women one-on-one and face-to-face.Women in the control group were not given any treatment other than routine care at family health centers. In routine care, pregnant women were subjected to edema, varicose veins, weight, blood pressure, pulse, laboratory findings, baby heart sounds, medication intake, chronic disease follow-up and vaccination. Pregnant women were provided with counseling if they had any questions. Postpartum women were subjected to blood pressure, fever, pulse, bleeding and laboratory findings follow-up and were provided with counseling if they had any questions.
  Interventions: Other: routine care

INTERVENTIONS:
Other: the psychoeducation intervention program booklet — Psychoeducation Program was composed of nine basic topics (postpartum period and care, adaptation to the role of motherhood and mother-infant bonding, postpartum psychological changes, frequency, causes, symptoms of PPD, effects on mother, child and community health, diagnosis and treatment, preventive practices, social support and suggestions for coping, breast milk and breastfeeding, breast care and practices, nutrition and baby care).
  Arms: intervention group
Other: routine care — routine care
  Arms: control group

SUMMARY:
This study was planned to evaluate the effects of psychoeducation intervention for postpartum care on postpartum depression and breastfeeding.

DETAILED DESCRIPTION:
The pregnant women included in the sample were informed about the study and their written informed consent was obtained. Six interviews were conducted with the pregnant women, four at one-week intervals before birth, and one on the tenth day and sixth week after birth. These interviews were conducted with the women one-on-one and face-to-face.Women in the control group were not given any treatment other than routine care at family health centers. The psychoeducation program was applied to the women in the intervention group in six interviews.

ELIGIBILITY:
Inclusion Criteria:

* 20-34. Women who are at the gestational age,
* over 18 years of age,
* planning to breastfeed,
* have no visual,
* hearing or mental disabilities,
* have a healthy fetus on ultrasonography

Exclusion Criteria:

* Women with depression and other mental illnesses diagnosed by a physician,
* those taking medication related to their mental illness,
* those who gave birth prematurely,
* those with contraindications to breastfeeding and newborns (head and spine anomalies such as anencephaly/spina bifida, having a fetus with brain anomalies such as hydrocephalus/microcephaly, active substance use or HIV diagnosis, etc.),
* those who were included in the study in the 3rd trimester but whose birth weight was less than 2500 grams,
* those whose babies were taken to the neonatal intensive care unit due to any postpartum complications and those who had premature babies (born before 37 weeks of gestation),
* those who did not participate in more than one interview

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Antenatal Breastfeeding Self-Efficacy Scale | 1 day (first meeting during pregnancy)
  The scale consists of a total of 20 items. The scale is a 5-point Likert type. The lowest score that can be obtained from the scale is 20 and the highest score is 100. An increase in the score obtained from the scale indicates that the perception of breastfeeding self-efficacy has increased.
Edinburgh Postpartum Depression Scale | 1 day (first meeting during pregnancy and at the sixth week postpartum)
  It is a 10-item self-report scale that measures maternal depressive symptoms over the past seven days. Higher scores reflect more depressive symptoms. Symptoms are rated on a 4-point Likert scale with scores ranging from 0 to 30. The cut-off score of the scale was determined as ≥13. If the total score of the scale is 12 or less, the participant is not at risk for PPD, but if he scores 13 or more, he is at risk.
Postpartum Breastfeeding Self-Efficacy | sixth week postpartum
  Breastfeeding Self-efficacy Short Form is a 5-point Likert-type scale. The lowest score that can be obtained from the scale is 14 and the highest score is 70. A higher score indicates higher breastfeeding self-efficacy.
Personal Information Form | 1 day (first meeting during pregnancy)
  The form created to determine the socio-demographic characteristics of the individuals included in the research was prepared by the researcher in line with the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Özhüner, Principal Investigator — Eskişehir Vadişehir Family center odunpazarı Turkey; nebahat özerdoğan, Study Director — Eskisehir Osmangazi University odunpazarı turkey
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozhuner Y, Ozerdogan N. The effect of psychoeducational intervention on postpartum care on postpartum depression and breastfeeding: a randomized controlled trial. BMC Nurs. 2025 Nov 26;24(1):1449. doi: 10.1186/s12912-025-04079-5. PMID 41299439